CLINICAL TRIAL: NCT05990244
Title: Comprehensive Assessment of Tumor Stiffness and Adhesion in Glioma Using Magnetic Resonance Elastography: A Prospective Study
Brief Title: Magnetic Resonance Elastography in Glioma: Exploring Tumor Stiffness and Adhesion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yu Shi, Deputy director of department of radology, Shengjing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ShengjingH_glioma2023
Record Dates: First submitted 2023-08-06; First posted 2023-08-14 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Glioma
Keywords: Magnetic Resonance Elastography; Brain tumor; Glioblastoma; MR elastography; Tumor molecular pathology
MeSH Terms: conditions — Glioma; Brain Neoplasms; Glioblastoma | interventions — Elasticity Imaging Techniques; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (MRE, tumor grade, tumor stiffness and adhesion) (Experimental): Patients undergo a preoperative routine MRI scan and MRE the day before their scheduled surgery to assess tumor stiffness and adhesion. Additionally, molecular pathological analysis will be performed to identify genetic alterations in gliomas. During surgery, the tumor stiffness and adhesion will be assessed and recorded by the surgeon according to established evaluation criteria.
  It is important to note that the surgeon does not have prior knowledge of the tumor's specific stiffness before the surgery. This information is typically obtained through intraoperative assessment and observation.
  Interventions: Diagnostic Test: Magnetic Resonance Elastography; Procedure: Assessment and Recording

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Elastography — Undergo MRE and routine MRI
  Other Names: MRE
Procedure: Assessment and Recording — Undergo recording of tumor stiffness during surgery and molecular pathological classification through genetic analysis

SUMMARY:
this study will investigate the relationship between tumor stiffness and adhesion in gliomas using MRE. By utilizing preoperative MRE and Intraoperative neuronavigation, followed by comprehensive molecular pathology analysis, we aim to explore the correlation of tumor stiffness and adhesion with molecular and genetic characteristics of gliomas. Additionally, the predictive value of MRE in terms of pathological staging and prognosis will be determined. This research may pave the way for improved clinical decision-making, personalized treatment approaches, and more accurate clinical trials for glioma patients.

DETAILED DESCRIPTION:
Magnetic Resonance Elastography (MRE) is an advanced imaging technique that measures the mechanical properties of tissues, providing valuable information about tissue stiffness, elasticity, and adhesion. In the case of gliomas, a type of brain tumor arising from glial cells, MRE has shown promising potential in the diagnosis, classification, and prediction of pathological and molecular features.

This clinical trial aims to investigate the relationship between tumor stiffness, adhesion, glioma grading, and genetic alterations by combining magnetic resonance elastography (MRE) imaging findings with molecular pathological analysis. Moreover, the study aims to predict patient survival based on the physical properties of the tumor.

Preoperatively, we will use MRE to enhance the accuracy of navigation and determine tumor stiffness and adhesion properties. Intraoperatively, under the guidance of neuronavigation, tissue samples will be obtained, and the operating surgeon will assess the tumor's stiffness, elasticity, and degree of adhesion.

Postoperatively, all tissue specimens will undergo molecular pathological analysis. The integration of MRE findings with molecular pathology data will enable precise classification and subtyping of gliomas.

Furthermore, all patients will receive systematic treatment after surgery, and long-term follow-ups will be conducted. This comprehensive approach combining MRE, molecular pathology analysis, and clinical follow-up aims to investigate the predictive value of MRE in terms of molecular pathological features and prognosis in gliomas.

ELIGIBILITY:
Inclusion Criteria:

1. age older than 18 years
2. Karnofsky performance status higher than 60
3. with written informed consent
4. MRE performed within one week before surgery
5. tumor diameter > 2 cm

Exclusion Criteria:

1. previous treatment for glioma
2. inability to complete MRE due to intolerance (e.g., vibration-related discomfort or claustrophobia)
3. completed MRE with suboptimal wave image quality (e.g., motion artifacts or inad-equate wave amplitude)
4. failure to proceed with surgery after MRE
5. missing IDH results

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Surgical assessment of tumor stiffness | Baseline to 6 weeks
  The surgeon will score the tumor stiffness in seven aspects, ranging from 1 to 5 points: Tumor size; Shape of tumor; Tumor texture; Stiffness of the tumor's capsule; Stiffness of the tumor's central region; Primary methods of tumor removal; Features of tumor's capsule.
Surgical assessment of tumor adhesion | Baseline to 6 weeks
  The surgeon will score the tumor's adhesion based on seven aspects, ranging from 1 to 4 points: Stripping instruments; Frequency of use of sharp instruments; Adhesion range; Degree of tumor resection; Cranial nerve anatomy preservation; Brain tissue anatomy preservation; Neurological function (compared with preoperative).
Radiological assessment of tumor stiffness | MRE performed within one week before surgery
  Tumor stiffness, measured in kilopascals (kPa), will be compared with its normal-appearing contralateral white matter using MRE by creating a lesion region of interest (ROI). Images were acquired on a 3T MR imaging unit with a vibration frequency of 60 Hz. The performance of the use of tumor stiffness to predict tumor grade was evaluated with the Wilcoxon rank sum, 1-way ANOVA, and Tukey-Kramer tests.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Shi, MD, Principal Investigator — Shengjing Hospital; Anhua Wu, MD, Principal Investigator — Shengjing Hospital; Wen Cheng, MD, Principal Investigator — Shengjing Hospital; Xiufang A( Ren, MD, Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murphy MC, Huston J 3rd, Glaser KJ, Manduca A, Meyer FB, Lanzino G, Morris JM, Felmlee JP, Ehman RL. Preoperative assessment of meningioma stiffness using magnetic resonance elastography. J Neurosurg. 2013 Mar;118(3):643-8. doi: 10.3171/2012.9.JNS12519. Epub 2012 Oct 19. PMID 23082888
- [Background] Hughes JD, Fattahi N, Van Gompel J, Arani A, Meyer F, Lanzino G, Link MJ, Ehman R, Huston J. Higher-Resolution Magnetic Resonance Elastography in Meningiomas to Determine Intratumoral Consistency. Neurosurgery. 2015 Oct;77(4):653-8; discussion 658-9. doi: 10.1227/NEU.0000000000000892. PMID 26197204
- [Background] Yin Z, Lu X, Cohen Cohen S, Sui Y, Manduca A, Van Gompel JJ, Ehman RL, Huston J 3rd. A new method for quantification and 3D visualization of brain tumor adhesion using slip interface imaging in patients with meningiomas. Eur Radiol. 2021 Aug;31(8):5554-5564. doi: 10.1007/s00330-021-07918-6. Epub 2021 Apr 14. PMID 33852045
- [Background] Yin Z, Hughes JD, Trzasko JD, Glaser KJ, Manduca A, Van Gompel J, Link MJ, Romano A, Ehman RL, Huston J 3rd. Slip interface imaging based on MR-elastography preoperatively predicts meningioma-brain adhesion. J Magn Reson Imaging. 2017 Oct;46(4):1007-1016. doi: 10.1002/jmri.25623. Epub 2017 Feb 14. PMID 28194925
- [Background] Pepin KM, McGee KP, Arani A, Lake DS, Glaser KJ, Manduca A, Parney IF, Ehman RL, Huston J 3rd. MR Elastography Analysis of Glioma Stiffness and IDH1-Mutation Status. AJNR Am J Neuroradiol. 2018 Jan;39(1):31-36. doi: 10.3174/ajnr.A5415. Epub 2017 Oct 26. PMID 29074637